CLINICAL TRIAL: NCT02762253
Title: Study of the Safety and Effectiveness of Photochemically Induced Collagen Cross-Linking at an Irrandiance of 18 mW/cm2 in Eyes With Keratoconus or Ectasia.
Brief Title: Study of the Safety and Effectiveness of Photochemically Induced Collagen Cross-Linking in Eyes With Keratoconus.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No IND submitted to the FDA
Sponsor: Nvision Laser Eye Centers (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NV001
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Riboflavin drops - epithelium on or off (Other): Riboflavin is applied with Epithelium on or with it off. 6 months follow up to find out magnitude of Decrease in Kmax
  Interventions: Drug: Riboflavin drops

INTERVENTIONS:
Drug: Riboflavin drops — Riboflavin drops were used every 2 minutes for 30 minutes on the cornea then exposed to 5 minutes of Ultraviolet light at an intensity of 18mW/cm2
  Other Names: Rincolin

SUMMARY:
This study is being conducted to assess the safety and effectiveness of photochemically induced collagen cross- linking (CCL) at irradiance of 18mW/cm2 in eyes with Keratoconus and Ecstasia.

DETAILED DESCRIPTION:
Riboflavin drops are used every 2 minutes for 30+ minutes until the corneal stroma is saturated with Riboflavin as evidenced by observing Riboflavin in the Anterior chamber. Two arms in the study, one uses Riboflavin with Epithelium on and the other with Epithelium off. Once it is observed that the Riboflavin has penetrated the stroma and is seen in the anterior chamber, the cornea is exposed to Ultraviolet light at an irradiance level of 18mW/cm2 for 5 minutes. A contact lens is applied until the epithelium has fully healed in 3 to 5 days. The study is for 6 months. The corneal curvature as well as the uncorrected and best corrected vision and corneal thickness are evaluated pre-operatively and at 6 months. The primary variable that is assessed to determine the efficacy of the drug is the Kmax - Steep corneal curvature. Secondary effectiveness criteria are uncorrected and best corrected vision and corneal thickness. adverse events are also monitored.

ELIGIBILITY:
INCLUSION CRITERIA GENERAL:

1. 12 years of age or older
2. Signed written informed consent
3. Willingness and ability to comply with schedule for follow-up visits
4. Contact lens removal prior to evaluation and treatment
5. Candidates must also have two of the following criteria:

   1. Presence of central or inferior steepening on the Pentacam or Orbscan map consistent with Keratoconus.
   2. Axial topography consistent with keratoconus.
   3. Steepest keratometry (Kmax) value of 47.00D

INCLUSION CRITERIA FOR ECTASIA:

History of having undergone a keratorefractive procedure and 2 of the following criteria:

1. Steepening by topography, either Pentacam or Orbscan
2. Thinning of cornea
3. Shift in the position of thinnest portion of cornea
4. Change in refraction with increasing myopia
5. Development of myopic astigmatism
6. Development of irregular astigmatism
7. Loss of BSCVA

   EXCLUSION CRITERIA:

   I. Eyes classified as either normal or atypical normal 2. Corneal pachymetry 350 microns at the thinnest point measured by Pentacam in the eye to be treated 3. A history of chemical injury or delayed epithelial healing in the eye to be treated.

   4. Pregnancy (including plan to become pregnant) or lactation during the course of the study 5. A known sensitivity to study medications 6. Patients with nystagmus or any other condition that would prevent a steady gaze during the treatment 7. Inability to cooperate with diagnostic tests. 8. Patients with a concomitant condition that, in the investigator's opinion, would interfere with or prolong epithelial healing.

   9. Taking Vitamin C (ascorbic acid) supplements within 1 week of the cross-linking treatment.

   10. Patients who are unable to remain supine and tolerate a lid speculum for an extended period of time.

   -

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2012-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Keratometry | 6 months
  The change in maximum keratometry (Kmax) from baseline will be evaluated at 6 months for all eyes. Data will be summarized using descriptive statistics.

SECONDARY OUTCOMES:
manifest refraction | 6 months
  The change in manifest refraction at 6 months compared to pre op
Visual Acuity | 6 months
  Change in BSCVA and UCVA compared to the baseline examination will be evaluated at 6 months postoperatively.
Central Pachymetry | 6 months
  The change in central pachymetry (as measured by Pentacam) from baseline will be evaluated at 6 months postoperatively. Data will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: tom s tooma, md, Principal Investigator — NVISION Eye Centers
Locations (11):
- United States (11):
  - NVISION Camarillo, Camarillo, California
  - NVISION Sacramento, Citrus Heights, California
  - NVISION Fullerton, Fullerton, California
  - NVISION Laguna Hills, Laguna Hills, California
  - NVISION Newport Beach, Newport Beach, California
  - NVISION Ontario, Ontario, California
  - NVISION La Jolla, San Diego, California
  - Berg Feinfield Vision Center, Sherman Oaks, California
  - NVISION Torrance, Torrance, California
  - NVISION Las Vegas, Las Vegas, Nevada
  - Teplick Custom Vision, Beaverton, Oregon

IPD SHARING:
Plan to Share IPD: Undecided